CLINICAL TRIAL: NCT00469846
Title: Supplementation With L-Arginine and Antioxidant Vitamins During Pregnancy in a Medical Food to Reduce the Risk of Preeclampsia in a High Risk Population
Brief Title: L-Arginine and Antioxidant Vitamins During Pregnancy to Reduce Preeclampsia
Acronym: L-Arg
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment and follow-up has been completed.
Sponsor: Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes (Other Government)
Collaborators: University of Pennsylvania (Other); Bill and Melinda Gates Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 212250-02071
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Last update posted 2007-05-08 (Estimated); Status verified 2007-04

CONDITIONS: Pre-Eclampsia
Keywords: Pre-Eclampsia; Hypertension,pregnancy-induced; Preterm labor
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Obstetric Labor, Premature | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: L-arginine supplementation in a medical food
Procedure: Vitamin C and E supplementation in a medical food

SUMMARY:
This study is intended to assess the efficacy of L-arginine supplementation with antioxidant vitamins delivered in a medical food in reducing the incidence of preeclampsia in a high-risk population.

DETAILED DESCRIPTION:
Preeclampsia is a syndrome of unknown origin characterized by hypertension, edema and proteinuria. It usually appears in the third trimester and occurs most frequently in primigravidas. Preeclampsia may be complicated by life-threatening conditions including seizures, severe hepatic dysfunction, renal failure and coagulopathy; it is one of the leading causes of maternal morbidity and mortality worldwide. Preeclampsia is cited as the leading cause of maternal death in surveys of maternal mortality in Mexico (25% of maternal deaths).

Specific Aim 1. To assess the efficacy of L-arginine supplementation with antioxidant vitamins delivered in a medical food in reducing the incidence of preeclampsia in a high-risk population. Two other groups will receive the food (bars) either with antioxidant vitamins alone or without vitamins in order to test the impact of vitamin supplements on prevention of preeclampsia. The primary hypothesis to be tested is that supplemental L-arginine in combination with antioxidant vitamins will significantly reduce preeclampsia (hypertension and proteinuria) and its complications in a high-risk population (women whose blood pressure is > 140/90 after 20 weeks gestation without proteinuria). Secondary hypotheses to be tested include that antioxidant vitamin supplementation contributes to the reduction in preeclampsia; that supplemental L-arginine and antioxidant vitamins will improve neonatal outcomes (reduced incidence of prematurity and intrauterine growth retardation); that preeclampsia is correlated inversely with plasma L-arginine levels, directly with the plasma levels of the endogenous NO synthase inhibitor, asymmetric dimethyl arginine (ADMA), and inversely with urinary NO metabolites, a marker of endogenous NO production; and that preeclampsia is inversely correlated with maternal plasma levels of antioxidant vitamins.

ELIGIBILITY:
Inclusion Criteria:

* Previous pregnancy complicated with pre-eclampsia/eclampsia
* Singleton pregnancy
* Gestational age >20 weeks <34 weeks
* Protein excretion < 300 mg/day

Exclusion Criteria:

* Multiple gestation
* Major fetal anomaly
* Pre-existing hypertension
* Pre-existing renal disease
* Diabetes
* Collagen vascular disease
* Cancer or strong family history of cancer in first degree relatives
* Preexisting maternal disease requiring medication

Ages: 19 Years to 32 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 585 (Actual)
Dates: Start 2001-01; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Development of preeclampsia | During pregnancy

SECONDARY OUTCOMES:
Development of eclampsia | During pregnancy
Occurrence of HELP syndrome | During pregnancy
Occurrence of preterm labor, preterm premature rupture of the membranes | During pregnancy
Gestational age at delivery | End of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Vadillo-Ortega, M.D.,Ph.D., Principal Investigator — Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes
Locations (2):
- Univesity of Pennsylvania, Philadelphia, Pennsylvania, United States
- Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes, Mexico City, D.F., Mexico

REFERENCES:
- [Derived] Vadillo-Ortega F, Perichart-Perera O, Espino S, Avila-Vergara MA, Ibarra I, Ahued R, Godines M, Parry S, Macones G, Strauss JF. Effect of supplementation during pregnancy with L-arginine and antioxidant vitamins in medical food on pre-eclampsia in high risk population: randomised controlled trial. BMJ. 2011 May 19;342:d2901. doi: 10.1136/bmj.d2901. PMID 21596735